CLINICAL TRIAL: NCT02894086
Title: A Retrospective Study of the Feasibility of Ambulatory Appendicectomy for Acute Appendicitis (Based on Data From the PMSI French National Hospital Information System) in the Adults Hospitalized Between December 2013 and December 2014
Acronym: PMSIApp
Status: Withdrawn | Type: Observational
Why Stopped: Investigator choice
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2015-35 Pr-REGIMBEAU-2
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Appendicitis
Keywords: acute appendicitis; ambulatory appendicectomy
MeSH Terms: conditions — Appendicitis | interventions — Database Management Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Other: database. — database

SUMMARY:
Acute appendicitis is a frequent surgical emergency, with an estimated incidence of about 80,000 cases a year (in France). It mainly affects young adults but is associated with a low complication rate and a short stay in hospital. Ambulatory treatment is an innovative type of care in which the patient is hospitalized for less than 12 hours and does not stay overnight in hospital.

Ambulatory care is based on the guidelines issued by three French learned societies (the SFCD, the ACHBT and the AFCA) and has been defined by the French government as a national priority.

The literature data show that 20% of patients undergoing appendicectomy for acute appendicitis can be treated on an ambulatory basis. However, the success factors for short-stay care (hospitalization <24 hours) or ambulatory care (hospitalization <12 hours) have yet to be identified.

The investigators thus intend to perform a retrospective study of data from the PMSI French national hospital information system, in order to identify factors that are predictive of a length of hospital stay below 24 hours in patients having undergone appendicectomy for acute appendicitis during 2013 in France. The objective is to define the population of patients that could potentially benefit from ambulatory care.

ELIGIBILITY:
Inclusion Criteria:

Medical criteria:

* Patients operated on for acute appendicitis between December 2013 and December 2014

Sociodemographic criteria:

* Adult patients (aged between 18 and 75, inclusive)
* Social security coverage

Exclusion Criteria:

Sociodemographic criteria:

* Patients under the age of 18
* Pregnancy or breastfeeding
* Legal guardianship or incarceration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated on for acute appendicitis between December 2013 and December 2014
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
identify the population of patients having been hospitalized for less than 24 hours. | during 1 year (from december 2013 to december 2014)
  The ICD-10 diagnostic codes for acute appendicitis, stored in the PMSI.

CONTACTS AND LOCATIONS:
Overall Officials: REGIMBEAU Jean-Marc, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France